CLINICAL TRIAL: NCT00003885
Title: Phase II Study of Arsenic Trioxide in Relapsed/Refractory Acute Leukemia and Blast Crisis of Chronic Myeloid Leukemia
Brief Title: Arsenic Trioxide in Treating Patients With Recurrent or Refractory Acute Leukemia, Chronic Myeloide Leukemia, Myelodysplasia, Lymphoma, or Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Our Lady of Mercy Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067053; OLMMC-9808; OLMMC-FDR001699; NCI-V99-1545
Record Dates: First submitted 1999-11-01; First posted 2004-08-18 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2000-06

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; blastic phase chronic myelogenous leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; previously treated myelodysplastic syndromes; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Lymphoma, T-Cell, Cutaneous; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have recurrent or refractory acute leukemia, chronic myeloid leukemia, myelodysplasia, lymphoma, or myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of arsenic trioxide on the remission rate in patients with recurrent or refractory acute leukemia, blast crisis chronic myeloid leukemia, myelodysplasia, lymphoma, or myeloma. II. Determine the time to progression and survival in patients treated with this regimen. III. Determine the toxic effects of this regimen in these patients.

OUTLINE: Patients are stratified into 1 of 8 categories: first relapse no greater than 6 months after complete response vs second relapse or refractory vs prior hematologic disorder vs myeloid blast crisis of chronic myeloid leukemia vs lymphoid leukemia vs lymphoma vs myeloma vs myelodysplasia. Patients receive IV arsenic trioxide over 2-3 hours for 5 consecutive days with 2 days of rest. Treatment continues in the absence of disease progression until complete response or 90 days is reached. Upon achieving complete response, treatment is discontinued for 30 days. Patients exhibiting complete response receive a second 28 day course of consolidation therapy while in remission starting no sooner than 31 days after the end of induction therapy. Patients are followed monthly.

PROJECTED ACCRUAL: A total of 14-29 patients per lymphoma and myeloma stratum and a total of 31 patients per leukemia stratum will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or refractory acute leukemia (myeloid or lymphoid), blast crisis chronic myeloid leukemia, myelodysplasia, lymphoma, or myeloma of all FAB subtypes

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 6 weeks Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL (except for leukemic infiltration dysfunction) Alkaline phosphatase less than 2 times upper limit of normal (except for leukemic infiltration dysfunction) Renal: Creatinine no greater than 2.0 mg/dL Other: No active infection Not pregnant Fertile patients must use effective contraception No history of seizure disorders

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 2 weeks since prior chemotherapy (except hydroxyurea) No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: No other concurrent investigational agents Concurrent antibiotic therapy allowed for stable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1997-11

CONTACTS AND LOCATIONS:
Overall Officials: Janice P. Dutcher, MD, Study Chair — Our Lady of Mercy Medical Center
Locations (1):
- Our Lady of Mercy Medical Center, The Bronx, New York, United States